CLINICAL TRIAL: NCT04049279
Title: Migration in Total Hip Arthroplasty with a Cemented BiMobile Cup: Better Stability with More Cement? (Be-Mobile)
Brief Title: Migration in Total Hip Arthroplasty with a Cemented BiMobile Cup: Better Stability with More Cement?
Acronym: Be-Mobile
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JointResearch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL64196.100.17
Record Dates: First submitted 2019-07-04; First posted 2019-08-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Total Hip Arthroplasty; Osteoarthritis, Hip
Keywords: primary total hip arthroplasty; RSA; cement; Dual mobility cup
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BiMobile standard cement (Active Comparator): 25 patients will receive a cemented THA with a BiMobile dual mobility cup, in a standard size after optimal reaming, resulting in a cement mantle of approximately 2mm.
  Interventions: Procedure: BiMobile standard cement
- BiMobile larger cement (Active Comparator): 25 patients will receive a cemented THA with a BiMobile dual mobility cup, in one size smaller than standard after optimal reaming, resulting in a cement mantle of approximately 4mm.
  Interventions: Procedure: BiMobile larger cement
- Avantage standard cement (Active Comparator): 25 patients will receive a cemented THA with an Avantage dual mobility cup, in a standard size after optimal reaming, resulting in a cement mantle of approximately 2mm.
  Interventions: Procedure: Avantage standard cement

INTERVENTIONS:
Procedure: BiMobile standard cement — BiMobile dual mobility cup, in a standard size after optimal reaming, resulting in a cement mantle of approximately 2mm.
  Arms: BiMobile standard cement
Procedure: BiMobile larger cement — BiMobile dual mobility cup, in one size smaller than standard after optimal reaming, resulting in a cement mantle of approximately 4mm.
  Arms: BiMobile larger cement
Procedure: Avantage standard cement — Avantage dual mobility cup, in a standard size after optimal reaming, resulting in a cement mantle of approximately 2mm.
  Arms: Avantage standard cement

SUMMARY:
Objective: The main objective of this study is to compare the (early) migration of the cemented BiMobile cup at two year post-surgery between two different cup sizes after standard optimal reaming, and consequently adjusting the cement mantle into circa 2 or 4 mm, in patients with a primary cemented total hip arthroplasty (THA). Additionally, the results of the BiMobile cup will be compared to the Avantage cup, which is placed with a standard cup size, resulting in a cement mantle of approximately 2 mm.

Study design: A prospective single centre blinded randomised controlled trial.

Study population: All patients who meet the criteria to undergo a cemented THA.

DETAILED DESCRIPTION:
Rationale: Total hip arthroplasty (THA) is a commonly performed surgery in patients with end-stage osteoarthritis (OA) of the hip. Although it is known as a successful procedure, (recurrent) dislocation after THA is a major problem and results in a deterioration in quality of life. Dislocation after THA is the number one cause of early revision surgery.

Dual-Mobility (DM) acetabular cups should provide more stability and biomechanically reduce the risk of (early) dislocation. Potential disadvantages of DM cups are increased liner wear, psoas impingement and loosening. This might result in more revision surgery at mid- and longer-term follow-up for the cemented cups. If the cemented fixation technique improves, this might diminish the disadvantages of more revisions due to loosening in cemented cups. High quality evidence guiding the best technique for cemented fixation is however lacking. The risk of implant loosening might be reduced by increasing the amount of cement used for cup fixation. It is currently unknown whether size of the implant, and thereby the amount of cement, affects stability and survival. To fill this gap in knowledge, this study will compare cup migration, as an indicator for loosening, in a new dual mobility cup (BiMobile, Waldemar Link GmbH & Co. KG, Hamburg, Germany), using a larger or smaller cup size (and thereby different amounts of cement: approximately 2mm or 4mm cement mantle). These results will also be compared with the Avantage cup (ZimmerBiomet), which is yet considered as a standard dual mobility cup in the Netherlands. Migration will be measured with Rontgen Stereophotogrammetry Analysis (RSA), which is currently the gold standard for measuring early migration and predicting long term survival. A relatively new and less intensive way to measure migration of prostheses is the use of computer tomography (CT) scans, however there is still little scientific evidence on how accurately this can be done. This study therefore also measures the accuracy with which migration is measured, between CT scans and RSA.

Objective: The main objective of this study is to compare the (early) migration of the cemented BiMobile cup at two year post-surgery between two different cup sizes after standard optimal reaming, and consequently adjusting the cement mantle into circa 2 or 4 mm, in patients with a primary cemented THA. Additionally, the results of the BiMobile cup will be compared to the Avantage cup, which is placed with a standard cup size, resulting in a cement mantle of approximately 2 mm.

Study design: A prospective single centre blinded randomised controlled trial.

Study population: At the outpatient clinic of OLVG, all patients who meet the criteria to undergo a cemented THA will be screened for the in- and exclusion criteria.

Intervention:

Group A: 25 patients will receive a cemented THA with a BiMobile dual mobility cup, in a standard size after optimal reaming, resulting in a cement mantle of approximately 2mm.

Group B: 25 patients will receive a cemented THA with a BiMobile dual mobility cup, in one size smaller than standard after optimal reaming, resulting in a cement mantle of approximately 4mm.

Group C: 25 patients will receive a cemented THA with an Avantage dual mobility cup, in a standard size after optimal reaming, resulting in a cement mantle of approximately 2mm.

Main study parameters/endpoints:

Migration of the acetabular cup at two year postoperative, measured with RSA and CT. RSA x-rays will be collected at discharge, 6 weeks, 6 months, 1 year and 2 years after surgery. CT scans will be collected at discharge and 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring an elective primary cemented THA.
* Male patient ≥70 years old and female patient ≥65 years old.
* Ability and willingness to follow instructions and to return for follow-up evaluations.
* The patient is able to understand the meaning of the study and is willing to sign informed consent.
* Understanding the Dutch language.

Exclusion Criteria:

* The patient is morbidly obese, defined as Body Mass Index (BMI) of ≥ 40.
* The patient is expected to need lower limb joint replacement for another joint within one year.
* The patient has a systemic or metabolic disorder leading to progressive bone deterioration.
* The patient has a deformity or disease located in other joints than the hip that needs surgery and that is limiting their ability to walk.
* The patient has an active or suspected latent infection in or around the hip joint.
* The patient's bone stock is compromised by a disease or infection which cannot provide adequate support and/or fixation to the prosthesis.
* The patient is unable or unwilling to sign informed consent for this study.
* The patient is deemed unsuitable for participation in the study based on the investigator's judgment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Migration of the acetabular cup | 2 years postoperative
  Migration of the acetabular cup, measured with rontgen stereophotogrammetry analysis (RSA).

SECONDARY OUTCOMES:
Migration of the acetabular cup | 6 weeks, 6 months and 1 year postoperative
  Migration of the acetabular cup, measured with rontgen stereophotogrammetry analysis (RSA).
Patient reported outcomes on physical functioning | prior to surgery, 6 months, 1 year, 2 years and 5 years after surgery
  Difference in patient reported outcomes on physical functioning following primary THA with a BiMobile cup with 2mm cement, compared to the BiMobile cup with 4mm cement and the Avantage cup, measured with the Hip disability and Osteoarthritis Outcome Score Physical Short form (HOOS-PS). Interval level scores from 0 (no difficulty) to 100 (extreme difficulty).
Patient reported outcomes on quality of life. | prior to surgery, 6 months, 1 year, 2 years and 5 years after surgery
  Difference in patient reported outcomes on quality of life, following primary THA with a BiMobile cup with 2mm cement, compared to the BiMobile cup with 4mm cement and the Avantage cup, measured with the EuroQol 5 Dimensions (EQ-5D). A higher score means a worse quality of life, a lower score means a better quality of life. For the visual analogue scale (part of the EQ-5D), the lowest means the worst an the highest score means the best health score.
Patient reported outcomes on pain | prior to surgery, 6 months, 1 year, 2 years and 5 years after surgery
  Difference in patient reported outcomes on pain, following primary THA with a BiMobile cup with 2mm cement, compared to the BiMobile cup with 4mm cement and the Avantage cup, measured with the Numeric Ratin Scale (NRS) for pain in rest and during weight bearing. 0 means no pain, 10 means the most extreme pain.
Patient Satisfaction | prior to surgery, 6 months, 1 year, 2 years and 5 years after surgery
  patient satisfaction will be scored with an anchor question about general daily functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Poolman, MD, PhD, Principal Investigator — OLVG
Locations (1):
- OLVG, Amsterdam, Netherlands